CLINICAL TRIAL: NCT07237646
Title: The Effect of Virtual Game Simulation and Virtual Reality-Based Learning Tool on Nursing Students' Thoracic and Lung Physical Examination Knowledge and Satisfaction: A Randomized Controlled Trial
Brief Title: Virtual Game Simulation and Virtual Reality-Based Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Yadigar Ordu, Associate Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Physical examination
Record Dates: First submitted 2025-09-27; First posted 2025-11-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Satisfaction, Personal; Knowledge
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: three groups (two interventions (virtual game simulation (Intervention-I) -virtual reality-based learning tool (Intervention-II)- one control)
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and evaluator blinding will be ensured in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual game simulation (Experimental): Students in this class will play the Virtual Game Simulation for Thorax and Lung Physical Examination located at https://nursinggames.net/tr/.
  Interventions: Other: Virtual game simulation
- Virtual reality-based learning tool (Experimental): Students in this class will experience the Thoracic and Lung Physical Examination featured in a virtual reality-based learning tool.
  Interventions: Other: Virtual reality-based learning tool
- Control (Active Comparator): Students in this class will learn Thoracic and Lung Physical Examination using traditional learning methods (theory, question and answer, discussion).
  Interventions: Other: Control

INTERVENTIONS:
Other: Virtual game simulation — The virtual game simulation was prepared for nursing students to learn thoracic and lung physical examination.
  Arms: Virtual game simulation
Other: Virtual reality-based learning tool — The virtual reality-based learning tool was designed for nursing students to experience thoracic and lung physical examination skills on a virtual patient in a life-like environment.
  Arms: Virtual reality-based learning tool
Other: Control — Traditional teaching method (question-answer, lecture, discussion) will be used.
  Arms: Control

SUMMARY:
The purpose of this study is to determine the effects of a virtual game simulation and a virtual reality-based learning tool on nursing students' knowledge and satisfaction with thoracic and lung physical examinations. Two different teaching methods involving technology will be used in the study. No studies have been found that have examined the thoracic and lung physical examination knowledge of nursing students using a virtual game simulation and a virtual reality-based student tool. The study will utilize a three-group (two interventions (virtual game simulation (Intervention-I) - virtual reality-based learning tool (Intervention-II) - one control) pretest-posttest randomized controlled trial design. The population will consist of 119 students enrolled in the second year of nursing at Gazi University Faculty of Nursing in the 2025-2026 Fall Semester and taking the elective course "Health Assessment" coded HEM 205. The sample will consist of 60 students (20 Intervention-I, 20 Intervention-II, 20 control) who met the inclusion criteria and agreed to participate in the study. Data will be collected using a "Descriptive Characteristics Form," a "Thoracic and Lung Physical Examination Knowledge Test," and a "Satisfaction with Education Methods Survey." First, all students will receive a one-hour theoretical training on thoracic and lung physical examination. Following the training, all students will receive a one-hour laboratory demonstration on thoracic and pulmonary physical examinations. All students will then be briefed, and a pretest will be administered the following week. The study will be implemented one week after the pretest. Students will be randomly assigned to three groups. The first group will play a virtual game simulation on thoracic and pulmonary physical examinations. The second group will experience a virtual reality-based learning tool. The third group, consisting of the control and excluded students, will be evaluated in a classroom environment using question-and-answer sessions. All students will then be informed that a posttest will be administered. The posttest will be administered one week later. After the posttest, all students will be provided with hands-on experience with technology-based learning methods.

DETAILED DESCRIPTION:
One of the teaching methods that incorporates technology in nursing education is virtual game simulation, a two-dimensional (2D) virtual computer game featuring simulated people that allows students to actively participate in a clinical scenario. Virtual game simulations are a pedagogical method that allows students to practice critical thinking and decision-making skills by using simulated patients in scenarios involving different clinical environments. Studies using virtual game simulations have been conducted with nursing students in the fields of obstetrics, pediatrics, geriatrics, mental health, surgery, respiratory diseases, emergency health, and the nursing process. These studies indicate that virtual game simulations increase students' knowledge, feedback, interaction, participation, self-confidence, self-efficacy, satisfaction, critical thinking, decision-making skills, learning, and psychomotor skills. This study is expected to make significant contributions to the literature by evaluating the effectiveness of providing thoracic and lung examination training to nursing students through virtual game simulation.

Virtual reality is another method that incorporates technology in nursing education. Virtual reality is the user's active interaction with a computer-generated world through realistic scenarios. Virtual reality technology offers students an active learning environment independent of time and space. Virtual reality technology offers students a safe, motivating learning experience, and providing physical assessment training on a virtual patient is seen as an efficient alternative that will make future healthcare professionals more competent and equipped. A limited number of studies teaching physical assessment skills using virtual reality-based learning tools have found that the emphasis is on teaching inspection and auscultation skills. This study is expected to contribute significantly to the literature by evaluating the effectiveness of virtual reality-based thoracic and lung examination training for nursing students. This study is the first to use two different and innovative learning technologies in teaching thoracic and pulmonary examinations to nursing students, a field that has received limited research. No studies have been found in the literature examining the effectiveness of virtual game simulation and virtual reality technology on nursing students' learning. Therefore, the study is unique in its field. Therefore, the results of this study are expected to provide important information regarding teaching thoracic and pulmonary physical examinations to nursing students and to improve student satisfaction with both learning methods.

ELIGIBILITY:
Inclusion Criteria:

* The student must be taking the HEM 205 "Health Assessment" course for the first time.
* Students must not have any eye conditions that affect depth perception, such as amblyopia (lazy eye), anisometropia (differences in refraction between the two eyes), or strabismus (crossed eyes).
* Students must have no problems speaking and understanding Turkish.
* They must be willing to participate in the research.

Exclusion Criteria:

* Having a high school, associate's degree, or bachelor's degree in a health-related field;
* Taking the HEM 205 "Health Assessment" course as a secondary course;
* Not attending the thoracic and lung physical examination theoretical course;
* Not participating in laboratory exercises;
* Not participating in one of the research steps (pre-test, virtual game simulation, virtual reality-based learning tool, post-test);
* Completing and/or incomplete data collection forms;
* Wanting to withdraw from the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-11-04 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Knowlegde | Up to 1 month
  Thorax and Lung Physical Examination Knowledge Test
Personal satisfaction | Up to 1 month
  Satisfaction Survey with Training Methods

CONTACTS AND LOCATIONS:
Overall Officials: Nurcan Çalışkan, PhD, Study Director — Gazi University Faculty of Nursing
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No